CLINICAL TRIAL: NCT00988871
Title: Comparison of the Central Venous Pressures Measured From the Peripherally Inserted Antecubital Central Catheters and the Internal Jugular Vein Central Catheters in Liver Transplantation Recipients
Brief Title: Comparison of Central Venous Pressures (CVPs) Measured From Peripherally Inserted Central Catheters (PICC) and CICC in Liver Transplantation Recipients
Acronym: PICC
Status: Completed | Type: Observational
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Jung-Yeon Yun MD, PhD / Title: Staff anesthesiologist, Department of Anesthesiology and pain medicine, Research institute and hospital, National cancer center, Republic of Korea
Other Study IDs: PICC1342
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Last update posted 2009-10-02 (Estimated); Status verified 2009-10

CONDITIONS: Patients Cannulated With Both PICC and CICC.; The Rapidly Fluctuating Hemodynamics During LT.
Keywords: PICC (peripherally inserted central venous catheter); CICC (centrally inserted central venous catheter; CVP (central venous pressure); LT (liver transplantation); agreement
MeSH Terms: interventions — Catheterization, Peripheral

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Liver transplantation (LT) recipients: LT recipients who had both PICC and CICC at the same time according to the LT protocol of our hospital
  Interventions: Device: PICC, CICC

INTERVENTIONS:
Device: PICC, CICC — PICC insertion, CICC (advanced venous access with pulmonary artery catheter) insertion

SUMMARY:
Background: Central venous pressure (CVP) monitoring from the peripherally inserted central venous catheter (PICC) has not often been used because of the higher inherent resistance of the PICC due to its longer length and narrower lumen. The objective of this study was to assess the reliability of the CVP measured from PICCs as a predictor of the CVP measured from CICCs in the setting of rapidly fluctuating hemodynamic conditions during liver transplantation.

DETAILED DESCRIPTION:
According to the protocol of LT in our hospital, a PICC is concomitantly inserted with the pulmonary artery catheter (PAC) and 9-Fr advanced venous access (AVA) catheter for the LT recipient at anesthetic induction. PAC and AVA catheter are usually removed on the second postoperative day, and instead the PICC is used for the postoperative infusion of prostaglandin E1 which is very irritable to small peripheral vein. So we fortunately had chance to measure the CVPs from both CICC and PICC simultaneously in the same patients.

Methods: We measured the CVPs from the CICC and the PICC simultaneously during each main surgical period of adult liver transplantation (preanhepatic, anhepatic, reperfusion, and neo-hepatic period). Data are presented as means ± standard deviation. Statistical analysis was performed using simple linear regression analysis to observe whether changes in the PICCP were paralleled by simultaneous changes in the CICCP. Bland-Altman analysis was used to determine the degree of agreement between the two devices. Analysis of variance was performed to study whether there were changes in the CVP agreement profiles in regard to the different time periods of LT. Differences were regarded as being statistically significant when p values were less than 0.05.

(This observational study has been completed already.)

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who had been scheduled for elective liver transplant surgery
* Patients who had been placed with both PICC and CICC at anesthetic induction

Exclusion Criteria:

* Failure to insert PICC

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients who had been scheduled for elective liver transplant surgery, and placed with both PICC and CICC.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2008-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
PICCP: CVP measured from peripherally inserted antecubital central catheters in liver transplantation recipients | every 10 minutes during the liver transplantation
CICCP: CVP from IJV central catheters in liver transplantation recipients | every 10 minutes during the liver transplantation

CONTACTS AND LOCATIONS:
Overall Officials: So-Hee Park, PhD, Study Director — Department of cancer registration and biostatistics branch, Research institute and hospital, National cancer center, Republic of Korea; Soon-Ae Lee, MD.PhD., Study Director — Department of Anesthesiology and pain medicine, Research institute and hospital, National cancer center, Republic of Korea
Locations (1):
- National Cancer Center, 323 Ilsan-ro, Ilsandong-gu, Goyang-si, Gyeonggi-do, South Korea

REFERENCES:
- [Result] Black IH, Blosser SA, Murray WB. Central venous pressure measurements: peripherally inserted catheters versus centrally inserted catheters. Crit Care Med. 2000 Dec;28(12):3833-6. doi: 10.1097/00003246-200012000-00014. PMID 11153622
- [Result] McLemore EC, Tessier DJ, Rady MY, Larson JS, Mueller JT, Stone WM, Fowl RJ, Patel BM. Intraoperative peripherally inserted central venous catheter central venous pressure monitoring in abdominal aortic aneurysm reconstruction. Ann Vasc Surg. 2006 Sep;20(5):577-81. doi: 10.1007/s10016-006-9108-x. Epub 2006 Jul 27. PMID 16871437